CLINICAL TRIAL: NCT07000994
Title: Dobutamine During Major Abdominal Surgery: A Randomized Pilot Trial (PUSH-1)
Brief Title: Dobutamine During Major Abdominal Surgery
Acronym: PUSH-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. Alina Bergholz, MD, University of Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-100915-BO-ff
Record Dates: First submitted 2025-05-14; First posted 2025-06-03 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Intraoperative Myocardial Depression
MeSH Terms: interventions — Dobutamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dobutamine administration (Experimental): In patient assigned to dobutamine administration, dobutamine (concentration: 5 mg mL-1) will be administered with an infusion rate of 3 µg kg-1 min-1 (ideal body weight).
  Dobutamine administration will start with the beginning of surgery and will end after the end of surgery (incision-to-suture). The treating anesthesiologist may increase or stop dobutamine administration if clinically indicated. Whenever dobutamine-induced tachycardia (defined as a heart rate ≥120 beats per minute) or new-onset cardiac arrhythmia is noted, dobutamine administration will be stopped. Restarting dobutamine administration is at the discretion of the treating anesthesiologist.
  Interventions: Drug: Dobutamine
- Routine care (Active Comparator): In patients assigned to routine care, intraoperative hemodynamic management will be in accordance with routine care.
  Interventions: Other: Routine care

INTERVENTIONS:
Drug: Dobutamine — In patient assigned to dobutamine administration, dobutamine (concentration: 5 mg mL-1) will be administered with an infusion rate of 3 µg kg-1 min-1 (ideal body weight).
  Arms: Dobutamine administration
Other: Routine care — In patients assigned to routine care, intraoperative hemodynamic management will be in accordance with routine care.
  Arms: Routine care

SUMMARY:
The PUSH-1 trial is a randomized, single-center pilot trial investigating whether dobutamine administration is feasible in patients having major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients ≥18 years scheduled for elective major abdominal surgery under general anesthesia (expected surgery duration ≥ 120 minutes)
* Planned continuous intraarterial blood pressure monitoring using an arterial catheter for clinical indications not related to the trial

Exclusion Criteria:

* Emergency surgery
* Liver or kidney transplantation surgery
* Status of post transplantation of kidney, liver, heart, or lung
* Pregnancy
* Heart rhythms other than sinus rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of dobutamine administration | During surgery (incision-to-suture)
  The primary outcome "feasibility of dobutamine administration" is defined as dobutamine administration during >70% of surgery duration in >80% of all patients.

SECONDARY OUTCOMES:
Arterial hypotension | During surgery (incision-to-suture)
  Time-weighted average mean arterial pressure below 65 mmHg [mmHg]
Stroke volume index | During surgery (incision-to-suture)
  Median stroke volume index [mL m-2]
Heart rate | During surgery (incision-to-suture)
  Median heart rate [beats per minute]
Cardiac index | During surgery (incision-to-suture)
  Median cardiac index during surgery [L min-1 m-2]
Norepinephrine amount | During surgery (incision-to-suture)
  Total amount of administered norepinephrine divided by body weight and surgical duration [µg kg-1 min-1]

OTHER OUTCOMES:
Severe tachyarrhythmias | During surgery (incision-to-suture)
  Incidence of severe tachyarrhythmias (severe tachycardia defined as a heart rate >120 beats per minute or new abnormal heart rhythms)
Blood loss | During surgery (incision-to-suture)
  Estimated blood loss [mL]
Amount of fluids | During surgery (incision-to-suture)
  Total amount of fluid administration divided by surgical duration [mL h-1]
Red blood cell transfusion | During surgery (incision-to-suture)
  Red blood cell transfusion requirements [units]
Urine output | During surgery (incision-to-suture)
  Total urine output divided by surgical duration [mL h-1]
Hospital length of stay | Assessed up to 3 months
  Hospital length of stay [days]
Rehospitalization | Within 30 days after surgery
  Rehospitalization within 30 days after surgery (assessed based on electronic health records and/or telephone interviews)
Postoperative complications | Within 30 days after surgery
  Incidence of postoperative complications (assessed based on electronic health records and/or telephone interviews): acute myocardial infarction, acute kidney injury, stroke, surgical site infection, sepsis, infection requiring antibiotic treatment, renal replacement therapy, non-fatal cardiac arrest, and death

CONTACTS AND LOCATIONS:
Overall Officials: Alina Bergholz, MD, Principal Investigator — University Medical Centre Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No